CLINICAL TRIAL: NCT01135238
Title: The Use of Adrenalectomy in Patients With Solitary Adrenal Gland Metastases
Brief Title: Adrenalectomy for Solitary Adrenal Gland Metastases
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Melanie L. Richards, M.D., Associate Professor of Surgery, Mayo Clinic
Other Study IDs: 09-007747
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Adrenal Gland Metastases; Adrenalectomy
Keywords: adrenalectomy; metastasis; morbidity; mortality; survival
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The adrenal glands are one of the most common organs involved in metastatic disease. Metastases are the second most common type of adrenal mass, second only to adenomas. It is a frequent finding during autopsy with a reported rate as high as 27% in patients with known primary malignancy. Although several studies have found an increased survival in patients who undergo resection of solitary adrenal metastases the indications for adrenalectomy in cases of metastatic adrenal tumor remain controversial. Collinson et al reported an increased survival in patients with melanoma. Median survival was 16 months for patients who underwent adrenalectomy compared to 5 months for patients with documented adrenal metastases treated non surgically.

The aim of this study is to compare retrospectively in case and control study, performing adrenalectomy, open or laparoscopic, versus supportive treatment for patients with solitary adrenal gland metastases. The investigators will review charts of patients between January 1994 and November 2009 who had adrenal gland metastases. The variables the inevstigators will compare are mortality, morbidity, primary tumour sites, histological cell type, age, tumour size, presence of synchronous metastases, mean time from diagnosis of primary tumor to treatment of adrenal metastases, indication for adrenalectomy, partial versus total adrenalectomy, suspected versus confirmed metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease to the adrenal gland

Exclusion Criteria:

* Primary adrenal neoplasm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing adrenalectomy for metastatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Adrenalectomy improves overall survival in patients with solitary metastasis | 25 years
  Survival data compared to historic controls

SECONDARY OUTCOMES:
Adrenalectomy can be performed with minimal morbidity in patients with metastatic lesions to the adrenal gland. | 25 years
  Operative outcomes compared to historic control patients undergoing adrenalectomy for non-maligant disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie L Richards, MD, Principal Investigator — Mayo Clinic